CLINICAL TRIAL: NCT06568666
Title: Comparision of Instant Effect of Lumbal and Sacroiliac Spinal Manipulation on Flexibility and Jumping Performance in Licensed Football Players
Brief Title: The Effect of Lumbar and Sacroiliac Manipulation on Football Players
Acronym: ELSMFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Assistant Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMT003
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Sports Physical Therapy; Neuromuscular Subluxation of Joint
Keywords: Spinal manipulation; Football; Flexibility; Vertical jump; Horizontal jump
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: The study involved 45 professional soccer players, divided into three groups: lumbar manipulation group (n=15), sacroiliac joint manipulation group (n=15), and control group (n=15). The manipulations were performed in a side-lying position, and tests (V - Sit Reach Test, horizontal and vertical jump tests) were performed 5 minute before manipulation techniques and after the manipulation techniques. Normal distribution parameters were determined using Kolmogorov-Smirnov and Shapiro Wilks tests. Quantitative data comparisons were made using Oneway Anova test, Tukey HDS test, Kruskal Wallis test, Dunn's test, Paired Sample T test, and Wilcoxon sign test. The p<0.05 level was used to determine statistically significant differences. The study used various tests to compare parameters, with the p<0.05 level being considered significant for statistically significant differences.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar manipulation group (Experimental): Lumbar spinal manipulation was also performed in the lateral recumbent position and HVLA thrust was applied to the segment where dysfunction was detected. The spinal process was determined as the contact point and the direction of HVLA thrust was from posterior to anterior.
  Interventions: Other: Lumbar spinal manipulation
- Sacroiliac Joint Manipulation Group (Experimental): The participant lies on his/her side on the healthy side; the lower knee is in extension while the upper knee is flexed and placed in the popliteal fossa of the lower knee. The participant's hands are left free on the ribs at the lower level. The practitioner crosses the movement barrier with the stabilizing hand, allowing the tissues to relax. The practitioner performs HVLA thrust of the iliac bone into posterior or anterior rotation (in the opposite direction of dysfunction) with the stabilizing hand.
  Interventions: Other: Sacroiliac joint manipulation
- Control Group (No Intervention): No treatment has been carried out.

INTERVENTIONS:
Other: Lumbar spinal manipulation — Lumbar spinal manipulation was performed in the lateral recumbent position and HVLA thrust was applied to the segment where dysfunction was detected. The spinal process was determined as the contact point and the direction of HVLA thrust was from posterior to anterior.
  Arms: Lumbar manipulation group
Other: Sacroiliac joint manipulation — The participant lies on his/her side on the healthy side; the lower knee is in extension while the upper knee is flexed and placed in the popliteal fossa of the lower knee. The participant's hands are left free on the ribs at the lower level. The practitioner crosses the movement barrier with the stabilizing hand, allowing the tissues to relax. The practitioner performs HVLA thrust of the iliac bone into posterior or anterior rotation (in the opposite direction of dysfunction) with the stabilizing hand
  Arms: Sacroiliac Joint Manipulation Group

SUMMARY:
The purpose of this study was to assess the immediate effects of chiropractic spinal manipulation methods on the lumbar and sacroiliac regions on professional soccer players' flexibility and leaping abilities.

DETAILED DESCRIPTION:
The study included 45 professional soccer players who were previously informed about the study and met the inclusion criteria. The 45 participants were then randomly divided into three groups: lumbar manipulation group (n=15), sacroiliac joint manipulation group (n=15) and control group (n=15).

The V-Sit Reach Test was used to assess flexibility, the vertical jump test (on the wall) was used to assess vertical jump, and horizontal jump was assessed with the help of a tape on the hall floor. Each test was repeated twice and the best result was recorded in centimeters (cm.). Five minutes after the initial tests were performed, the lumbar spinal manipulation group underwent lumbar spinal manipulation on the identified dysfunctional segment, the sacroiliac joint manipulation group underwent sacroiliac joint manipulation on the dysfunctional side, and the control group did not receive any treatment.

The same tests were then repeated without any waiting period and the best result was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Signing the voluntary consent form
* Being a male
* Being between ages of 18 - 35
* Playing professional soccer for a minimum of 6 months
* Asymptomatic dysfunction of the lumbar spine or sacroiliac joint.

Exclusion Criteria:

* Having an injury in the lower extremities
* Lumbar spine and sacroiliac region in the last 6 months
* Having a contraendication to the chiropractic treatments

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
V-Sit Reach Test | This test was performed 5 minutes before and immediately after the manipulation.
  The participant is advised to sit on the floor with his legs straight front. The toes are pointed up, the heels are in touch with the ground, and there is about a 30-centimeter distance between them. A line is drawn connecting the spots where the heels strike the ground, and this line is used as the zero line for measurements. The patient is urged to reach forward with his hands as far as he can while keeping his knees extended. The distance between the attained point and the zero point is measured in centimeters. The numerical value is preceded by (+) and (-), which denote the location relative to the zero point. The knees should be kept in extension during the test. To obtain a measurement result, the tested person repeats the movement twice and the practitioner records the best result (+) or (-) in cm.
Vertical Jump | This test was performed 5 minutes before and immediately after the manipulation.
  The athlete stands facing the platform allocated for the test. With one arm, he/she reaches the highest point possible, and the test administrator marks the platform. The athlete jumps and touches the highest place he or she is able to reach, and is then noted. The test administrator measures the distance between these two spots and notes it in centimeters. The test must be taken twice. The best results are considered.
Horizontal Jump | This test was performed 5 minutes before and immediately after the manipulation.
  It is a test that assesses athletes' balance, jumping strength, and lower extremity strength in both vertical and horizontal planes. The test starting location is marked on the floor with a marker. In this stance, the individual being tested waits for the required acceleration. They leap as far as possible utilizing their single and double legs, as directed by the test administrator. The distance from the starting position to the leap point is measured. The test is repeated twice, and the best result is recorded in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA HAKTAN HATIK, Study Director — Sinop University
Locations (1):
- Sefa Haktan Haktik, Sinop, Turkey (Türkiye)